CLINICAL TRIAL: NCT05375786
Title: Epidemiological Study on Asymptomatic Infections and Mild Illness With Covid-19 in Shanghai
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SCAM2022
Record Dates: First submitted 2022-05-13; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 infections: * SARS-Cov-2 RNA positive
  * without symptom or with mild clinical manifestations
  Interventions: Biological: Vaccination completion status

INTERVENTIONS:
Biological: Vaccination completion status — the relation between vaccination completion status and the target population

SUMMARY:
this study is to clarify the epidemiological characteristics of Omicron variant infected persons in Shanghai, such as distribution characteristics, host and clinical characteristics, disease outcome and risk factors. especially asymptomatic infections.

ELIGIBILITY:
Inclusion Criteria:

* SARS-Cov-2 RNA positive.
* asymptomatic or mild clinical manifestation.
* informed consent signed.

Exclusion Criteria:

* informed consent rejected.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Asymptomatic infections or mild Illness with covid-19 in fangcang shelter hospitals in Shanghai
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-04-02 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Viral clearance time | 2 months
  time from viral RNA positive to negative

CONTACTS AND LOCATIONS:
Overall Officials: Erzhen CHEN, Ph D, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data are not publicly available due to the privacy and ethical restrictions.